CLINICAL TRIAL: NCT03480659
Title: Breast Cancer Screening Using DNA Methylation Changes in Circulated Tumor, PBMC and T-cells DNA.
Brief Title: Detection of Breast Cancer With Non-invasive Method Based on DNA Methylation of Circulated Tumor DNA, PBMC
Status: Terminated | Type: Observational
Why Stopped: Experienced technical issues with plasma blood samples collected from patients.
Sponsor: HKGepitherapeutics (Industry)
Collaborators: Kazakh Research Institute of Oncology & Radiology (Other); Montreal EpiTerapia Inc. (Industry); Canada-Kazakhstan EpiTerapia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HKG-KZ-BrCa-101
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Breast Cancer Female
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA extracted from plasma and PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer: Early stage luminal A and triple negative breast cancer [TNBC] (estrogen receptor-negative (ER-), progesterone receptor-negative (PR-) and HER2-negative (HER2-)
- Control: Age matched control females

SUMMARY:
A central challenge in the fight against breast cancer is how to detect disease in a noninvasive manner before it is detectable by imaging methods. Although inroads have been made with more sensitive imaging techniques for earlier detection of breast cancer, these techniques are limited by the size of lesion that could be detected. Alternatively, several blood proteomic biomarkers have been proposed but none offer as of yet sufficient predictive power. Consequently, effective non-invasive tools as prognostic indicators and biomarkers of breast cancer are urgently needed.

The purpose of this study is to develop and test non-invasive biomarkers based on methylation changes in PBMC and circulated tumor DNA in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed breast cancer subtypes (DCIS and invasive)

Exclusion Criteria:

* Pregnant women
* Minors (subjects less than 18 years of age)
* Prisoners
* Patients with known infectious disease, such as human immunodeficiency virus (HIV), tuberculosis (TB), or hepatitis B, C
* Patients having other than one cancer
* Subjects unable to consent for themselves

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer females
Study Population: Patients will be assigned an ID that will be kept confidential according to hospital regulations. IDs will be randomized so that identity will not be revealed except to the approved hospital personnel. Methylation data will be returned to the hospital for follow up of progression of disease and for assessing early prediction of progression of Breast cancer and will be entered into the data base. Other clinical follow up data will be entered into the electronic data base. All data will be captured in case report form
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
DNA methylation of circulated tumor and PBMC DNA and its Correlation to Development and prediction of breast cancer | 6 months to 1 year
  We will develop the linear model and a threshold value differentiating breast cancer from control based on the 100 patient training set. The model will be provided to the researchers:
  Methylation score=CG1*b1+CG2*b2+ CG3*b3 + e
  CG1 is the methylation value of the first CG b1 is the regression coefficient for the first CG and e equals the intercept.
  We will develop the regression coefficient and intercept as well as the DNA methylation values for each patient for each CG. We will first compute the polygenic methylation score for each patient. Then based on the computer threshold based on the training cohort will call the samples as breast cancer or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Kazakh Institute of Oncology and Radiology, Almaty, Kazakhstan